CLINICAL TRIAL: NCT07279636
Title: A Randomized, Double-blind, Placebo-Controlled, Dose-Escalation, Phase Ia Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Oral Administration of Alpha-0261 Tablets in Adult Healthy Participants
Brief Title: A Study to Evaluate Single Doses of Alpha-0261 in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AlphaMol Science Ltd. (Shanghai) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Alpha-0261-001
Record Dates: First submitted 2025-11-29; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental)
  Interventions: Drug: Alpha-0261
- Single Ascending Dose (placebo) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alpha-0261 — Oral, tablet
  Arms: Single Ascending Dose
Other: Placebo — Oral, tablet
  Arms: Single Ascending Dose (placebo)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of Alpha-0261 tablets after single oral administration in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 and ≤ 55, male or female
* Weight: ≥ 50 kg for males, ≥ 45 kg for females; 19 kg/m2 ≤ body mass index (BMI) ≤ 28 kg/m2
* In general good health

Exclusion Criteria:

* Have a history of any severe allergic reaction or anaphylaxis
* Any condition, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol
* Have clinically significant abnormalities on clinical laboratory results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events | From enrollment to end of follow-up visit, up to approximately 1 week

SECONDARY OUTCOMES:
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Maximum Plasma Concentration (Cmax)
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Elimination half life (T 1/2)
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Area Under the Concentration-time Curve (AUC)
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Time to Reach The Maximum Plasma Concentration (Tmax)
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Apparent Systemic Clearance (CL/F)
Plasma PK of Alpha-0261 after single dose | From enrollment to end of treatment period, up to approximately 7 days
  Apparent Volume of Distribution (Vz/F)

CONTACTS AND LOCATIONS:
Locations (1):
- Bishan Hospital of Chongqing, Chongqing, China